CLINICAL TRIAL: NCT06765538
Title: Video Versus Face-to-face Preoperative Anaesthetic Assessment: a Randomized Clinical Trial on Safety and User Satisfaction
Brief Title: Video Versus Face-to-face Preoperative Anaesthetic Assessment
Acronym: VIDFACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Katrine Bredahl Buggeskov, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-24006615
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia; Telemedicine
Keywords: anaesthetic preassessment; telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video consultation (Experimental): Patients receiving video consultations
  Interventions: Other: Video consultation
- Physical consultation (No Intervention): Patients receiving physical consultations (standard care)

INTERVENTIONS:
Other: Video consultation — Preanaesthetic videoconsultation
  Arms: Video consultation

SUMMARY:
Randomized clinical trial rewieving difference between anaesthetic preassessment in physical consultations vs. video consultations.

DETAILED DESCRIPTION:
Preoperative anaesthetic assessment aims to reduce morbidity and mortality and are currently accepted as the gold standard of care for elective surgery. Technical advances in society have led to explora-tions within the telemedicine area which continues providing safe and effective services. The video versus face-to-face preoperative anaesthetic assessment (VIDFACE) trial aims to compare videobased preoperative anaesthetic assessment to standard face-to-face consultations with focus on patient safety and satisfaction including possible beneficial eco and economical effects compared to standard face-to-face consultations.

This is a randomised, single-centre, two-arm, assessor, and data analyst blinded clinical trial. We will enrol 2260 participants undergoing elective Ear-Nose-Throat or Tooth-Mouth-Jaw surgery. Participants will be randomised 1:1 stratified by malignant versus benign surgery to either video based preoperative anaesthetic assessment or face-to-face consultation. Data will be analysed by two blinded statisticians, and we will write abstracts covering all possible combinations of conclusions, before breaking the blind.

Results:

The primary outcome is the incidence of six predefined serious adverse events (SAE). Secondary outcomes are the proportion of participant with a change in anaesthesia plan as well as delays or cancellations on the day of surgery and patient satisfaction.

The VIDFACE trial will contribute valuable knowledge on the efficacy and safety on using video consultations in the an-aesthetic preoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

* ENT and TMJ patients
* Adults > 18 years
* Informed consent obtained after a consideration period of minimum 24 hours

Exclusion Criteria:

* If a patient is assessed unsuitable for the video technology in example, patients with severe mental challenges (dementia, retardation, etc.), they will not be included in the trial. If excluded, the patient receives standard care, face-to-face preoperative anaesthetic assessment.
* Local protocol screen patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2260 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
SAE | 30 day follow up
  All-cause mortality, all-cause admission to intensive care unit, bleeding requiring transfusion, infection requiring antibiotics, hospital readmission or prolonged hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosholdt SA, Denneborg MKG, Rosenkrantz O, Moller MH, Jakobsen JC, Olsen MH, Mogelmose A, Hesselfeldt RT, Buggeskov KB. Video Versus Face-To-Face Preoperative Anaesthetic Assessment: The VIDFACE Trial-A Statistical Analysis Plan. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70068. doi: 10.1111/aas.70068. PMID 40467292